CLINICAL TRIAL: NCT05500261
Title: The Anxiolytic Effect of Intranasal Dexmedetomidine for Severely Anxious Patients in Dental Treatments
Brief Title: Intranasal Dexmedetomidine for Severe Dental Anxiety: a Randomized Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SYSKY-2022-119-03
Record Dates: First submitted 2022-08-02; First posted 2022-08-15 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-07

CONDITIONS: Dental Anxiety
Keywords: Dexmedetomidine; Intranasal; Randomized controlled trial
MeSH Terms: interventions — Dexmedetomidine; Randomized Controlled Trials as Topic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 0.8 μg/kg intranasal dexmedetomidine (Experimental): Intranasal administration of 0.8 μg/kg dexmedetomidine
  Interventions: Drug: Dexmedetomidine
- 1.5 μg/kg intranasal dexmedetomidine (Experimental): Intranasal administration of 1.5 μg/kg dexmedetomidine
  Interventions: Drug: Dexmedetomidine
- 2.0 μg/kg intranasal dexmedetomidine (Experimental): Intranasal administration of 2.0 μg/kg dexmedetomidine
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — intranasal administration of dexmedetomidine
  Other Names: intranasal, randomized controlled trial, dental anxiety

SUMMARY:
Patients with dental anxiety only develop anxiety and fear about dental treatments. Patients with severe dental anxiety have difficulty cooperating with dental treatments, and can only complete dental treatments through general anesthesia, or even abandon treatments. Dexmedetomidine is a potent, highly selective α2-adrenoceptor agonist, which provides good anxiolytic, sedative and analgesic effects and is commonly used in anesthesiology and intensive care medicine departments, routinely intravenously. In recent years, intranasal administration of dexmedetomidine has also been reported for pediatric dentistry and adult alveolar surgery, showing good sedative and analgesic effects. However, these studies have problems such as single surgical types, small sample size, and few indicators analyzed. Therefore, the evaluation of intranasal administration of dexmedetomidine is still not comprehensive enough. Besides, the anxiolytic effect of dexmedetomidine for dental anxiety has not been reported yet. This project plans to carry out a randomized, double-blinded, placebo-controlled, two-stage clinical trial. We will firstly explore a reasonable dose, and secondly verify it with placebo as the control. We plan to measure the object indicators, including the NTI value, plasma cortisol, interleukin-6, blood pressure and heart rate, and to assess the subjective indicators using scales and questionnaires, thus comprehensively evaluating the effectiveness, safety and feasibility of the anxiolytic effect of intranasal dexmedetomidine for severe dental anxious patients, and preliminary exploring its mechanism additionally. We intend to help severe dental anxious patients completing dental treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Fully understand the purpose and significance of this trial, voluntarily participate in this clinical trial, and voluntarily sign an informed consent form;
2. Age 18 to 65 years old, regardless of gender;
3. Diagnosed by a dentist and needs dental treatment;
4. Can be immediately arranged for dental treatment after being evaluated by the clinician as having no contraindications;
5. Graded as severe dental anxious (obtained using the MDAS modified dental anxiety scale);
6. After controlling the symptoms of infection if with symptoms of acute/systemic infection, and can be arranged immediately after meeting the indications for dental treatments;
7. BMI is 18.5 kg/m2~25 kg/m2;
8. After resting for 30 min, the SBP < 180 mmHg, the DBP < 110 mmHg, and the 60≤HR ≤ 120 bpm;
9. For women who have not been menopausal or who have been under 1 year of menopause, a pregnancy test (blood or urine pregnancy test) should be performed during the screening period, and then the study and administration should be carried out after the pregnancy test is negative during the screening period.

Exclusion Criteria:

1. Subjects who are not considered by the researcher to be suitable for nasal drops (such as severe rhinitis, nasal malformations, etc.);
2. Subjects with a history of severe arrhythmias such as type II or above AV block or a history of cardiac insufficiency;
3. Subjects with a history of myocardial infarction or unstable angina in the 6 months before the screening period;
4. Subjects with a history of ischemic stroke or transient ischemic attack (TIA);
5. Subjects with poor blood pressure control after drug therapy (hypertension: SBP≥180 mmHg, and/or DBP≥110 mmHg, or hypotension: SBP <90 mmHg and/or DBP≤50 mmHg);
6. Subjects with psychiatric disorders (such as schizophrenia, anxiety, depression, etc.) and cognitive dysfunction, or have a history of epilepsy, or previous abuse of psychotropic drugs and narcotic drugs;
7. Subjects with a history of difficult airway disease or possibility, such as obstructive sleep apnea syndrome;
8. Randomly, within 1 year of random, a history of drug abuse, a history of drug abuse and a history of alcohol abuse, i.e., a subject who drank more than 2 units of alcohol per day on average (1 unit = 360 ml of beer or 45 ml of liquor or 150 ml of wine with an alcohol content of 40%);
9. Subjects who received selective alpha2-adrenoceptor agonists or antagonists within 14 days of randomization;
10. Those who are allergic to dexmedetomidine hydrochloride or items used in stomatology;
11. Pregnant or nursing women;
12. Those who have a birth plan within 30 days before the screening period and half a year after the end of the trial, and are unwilling or unable to take effective contraception measures;
13. Other circumstances in which the investigator determines that the subject is not suitable to participate in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2023-07-23 (Estimated); Study Completion 2023-07-23 (Estimated)

PRIMARY OUTCOMES:
Change of MDAS score | Change from baseline MDAS score right after finishing dental treatments, an average of 30 minutes
  Dental anxious score will be accessed by modified dental anxiety scale (MDAS), and the change of MDAS score will be calculated as the scores right after dental treatments minus the initial score before intervention.

SECONDARY OUTCOMES:
Change of plasma cortisol concentration | Change from baseline plasma cortisol concentration right after finishing dental treatments, an average of 30 minutes
  The change of plasma cortisol concentration will be calculated as the values right after dental treatments minus the initial values before intervention.
Change of NTI score | Change from baseline NTI score right after finishing dental treatments, an average of 30 minutes
  The depth of sedation will be accessed by NTI score using Narcotrend, and the change of NTI score will be calculated as the score right after dental treatments minus the initial score before intervention.
Change of OAA/S score | Change from baseline OAA/S score right after finishing dental treatments, an average of 30 minutes
  OAA/S score will be accessed by observer's assessment of alertness/sedation scale (OAA/S), which also represent the depth of sedation, and the change of OAA/S score will be calculated as the score right after dental treatments minus the initial score before intervention.
Change of blood pressure (BP) | Change from baseline BP right after finishing dental treatments, an average of 30 minutes.
  BP will be continuously accessed using an electrocardiogram monitor throughout the whole clinical process. BP value will be converted into mean arterial pressure (MAP) for comparison using the formula: MAP = (SBP + 2 × DBP)/3. Then the change of BP was presented as ΔMAP, which was calculated as the MAP at the point with the highest SBP minus the initial MAP right before the procedure.
Change of heart rate (HR) | Change from baseline HR right after finishing dental treatments, an average of 30 minutes.
  HR will be continuously accessed using an electrocardiogram monitor throughout the whole clinical process. Change of HR equaled the corresponding HR of the highest SBP subtracted by the initial HR.
Pain score | Through the completion of dental treatments, an average of 30 minutes.
  Pain score will be obtained via visual analogue scale (MDAS) for the subject to fill.
Percentage of thinking feasible of intranasal dexmedetomidine by participants | Through the completion of dental treatments, an average of 30 minutes.
  The feasibility of intranasal dexmedetomidine will be assessed through semistructured questionnaires. Items includes the reasons for nonparticipation; the acceptability of the trial and intranasal dexmedetomidine to participants; and the experience of the patients, the clinician performing the procedure, and the nursing staff taking care for patients during the study. The patients and clinic staffs filled the questionnaires right after the extraction process under our instruction. The outcome of the questionnaires was analyzed through counting and reported as a percentage (%).

CONTACTS AND LOCATIONS:
Overall Officials: Zeman Qin, Master, Principal Investigator — Department of General Dentistry, Sun Yat-sen Memorial Hospital, Sun Yat-sen University

IPD SHARING:
Plan to Share IPD: Yes
All of the data will be shared after publication of the paper of this trial
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will become available after the publication of the paper about this trial
Access Criteria: IPD will be accessed by the Data and Safety Monitoring Committee and all researchers in related fields
URL: http://www.medresman.org.cn

REFERENCES:
- [Background] Uusalo P, Guillaume S, Siren S, Manner T, Vilo S, Scheinin M, Saari TI. Pharmacokinetics and Sedative Effects of Intranasal Dexmedetomidine in Ambulatory Pediatric Patients. Anesth Analg. 2020 Apr;130(4):949-957. doi: 10.1213/ANE.0000000000004264. PMID 31206433
- [Background] Yoo H, Iirola T, Vilo S, Manner T, Aantaa R, Lahtinen M, Scheinin M, Olkkola KT, Jusko WJ. Mechanism-based population pharmacokinetic and pharmacodynamic modeling of intravenous and intranasal dexmedetomidine in healthy subjects. Eur J Clin Pharmacol. 2015 Oct;71(10):1197-207. doi: 10.1007/s00228-015-1913-0. Epub 2015 Aug 2. PMID 26233335
- [Background] Coursin DB, Coursin DB, Maccioli GA. Dexmedetomidine. Curr Opin Crit Care. 2001 Aug;7(4):221-6. doi: 10.1097/00075198-200108000-00002. PMID 11571417
- [Result] Shetty SK, Aggarwal G. Efficacy of Intranasal Dexmedetomidine for Conscious Sedation in Patients Undergoing Surgical Removal of Impacted Third Molar: A Double-Blind Split Mouth Study. J Maxillofac Oral Surg. 2016 Dec;15(4):512-516. doi: 10.1007/s12663-016-0889-3. Epub 2016 Apr 21. PMID 27833345
- [Result] Nooh N, Sheta SA, Abdullah WA, Abdelhalim AA. Intranasal atomized dexmedetomidine for sedation during third molar extraction. Int J Oral Maxillofac Surg. 2013 Jul;42(7):857-62. doi: 10.1016/j.ijom.2013.02.003. Epub 2013 Mar 14. PMID 23497981
- [Result] Cheung CW, Ng KF, Liu J, Yuen MY, Ho MH, Irwin MG. Analgesic and sedative effects of intranasal dexmedetomidine in third molar surgery under local anaesthesia. Br J Anaesth. 2011 Sep;107(3):430-7. doi: 10.1093/bja/aer164. Epub 2011 Jun 16. PMID 21685111
- [Result] Liu S, Wang Y, Zhu Y, Yu T, Zhao H. Safety and sedative effect of intranasal dexmedetomidine in mandibular third molar surgery: a systematic review and meta-analysis. Drug Des Devel Ther. 2019 Apr 23;13:1301-1310. doi: 10.2147/DDDT.S194894. eCollection 2019. PMID 31114165
- [Result] Ryu DS, Lee DW, Choi SC, Oh IH. Sedation Protocol Using Dexmedetomidine for Third Molar Extraction. J Oral Maxillofac Surg. 2016 May;74(5):926.e1-7. doi: 10.1016/j.joms.2015.12.021. Epub 2016 Jan 7. PMID 26850877